CLINICAL TRIAL: NCT02267967
Title: A Multi-Center, Open-Label, Phase Ib/II Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Sufatinib in Treating Advanced Neuroendocrine Tumors
Brief Title: Phase Ib/II Study of Sulfatinib in Treating Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-012-00CH1
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulfatinib (Experimental): Sulfatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle.
  Interventions: Drug: Sulfatinib

INTERVENTIONS:
Drug: Sulfatinib — Sulfatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle.
  Other Names: HMPL-012; Surufatinib

SUMMARY:
a multicenter, open-label phase Ib study to determine the safety, tolerability and preliminary efficacy of Sulfatinib 300 mg once a day in treating advanced neuroendocrine tumors

DETAILED DESCRIPTION:
The study population is patients with low- or intermediate-grade (G1 or G2) advanced NET who have failed in standard treatment or are unable to receive standard treatment.Sulfatinib 300 mg once a day (QD) will be orally administrated on a 28-day cycle. Investigators will evaluate the clinical tumor response to Sulfatinib, and if investigators determine that the patient can benefit from the continuation of treatment, the patient will continue the Sulfatinib treatment. The duration of study will be 2 years. At the time of study completion, if investigators believe patients can continue to benefit from the investigational product, patients may be provided with Sulfatinib with the agreement of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Be at least 18 years old;
3. Have a confirmed histological or cytological diagnosis of low- or intermediate-grade advanced NETs (unresectable or metastatic), for which standard treatment has failed or cannot be received. The NETs must meet the following criteria: (a) be GEP-NETs or NETs with the primary lesion located in tissue other than the lung or thymus (including unknown primary lesion location), with a mitotic count of ≤ 20/10 High Power Field [HPF] and a Ki67 index of ≤ 20%; or (b) be NETs of the lung or thymus (carcinoid) with a mitotic count of ≤ 10/10 High Power Field [HPF])
4. Have measurable lesions (according to RECIST 1.1);
5. Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale;
6. Have expected survival of more than 12 weeks;
7. Female patients with reproductive potential must agree to use an effective contraceptive method, for example, double-barrier device, condom, oral or injection birth control medication or intrauterine device, during the study and for 90 days after study completion.

Exclusion Criteria:

1. Absolute neutrophil count (ANC) of < 1.5×109/L, or platelet count of < 100 ×109/L, or hemoglobin < 9 g/dL;
2. Serum total bilirubin > 1.5 times the upper limit of normal (ULN);
3. ALT, AST or ALP > 2.5 ULN without hepatic metastases or ALT, AST or ALP > 5 ULN with hepatic metastases
4. Clinically significant serum potassium (regardless of potassium agent supplementation); serum calcium (ionic or binding to albumin post-adjusted) or clinically significant abnormal serum magnesium (regardless of magnesium agent supplementation);
5. Serum creatinine > 1.5 ULN (with the exception of CCR ≥ 60 ml/min based on 24-hour urine collection);
6. Urine protein > 2+, or 24-hour urine protein quantity >1 gram;
7. Uncontrolled hypertension, defined as: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90mmHg;
8. International Normalized Ratio (INR) > 1.5 ULN or activated partial thromboplastin time (aPTT) > 1.5 ULN. INR is only for patients not receiving anticoagulant therapy;
9. History or presence of digestive tract diseases, including active gastric/duodenal ulcer or ulcerative colitis, or active hemorrhage of an unresected gastrointestinal tumor, or an evaluation by investigators of having any other condition that could possibly result in gastrointestinal tract hemorrhage or perforation;
10. History or presence of serious hemorrhage (> 30 ml within 3 months), hemoptysis (> 5 ml fresh blood within 4 weeks) or a thromboembolic event (including transient ischemic attack) within 12 months;
11. Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrolment, severe/unstable angina pectoris or coronary artery bypass grafting, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment or left ventricular ejection fraction (LVEF) < 50%;
12. Other malignancies within the previous 5 years, with the exception of basal cell carcinoma, squamous-cell carcinoma post radical resection, or cervical carcinoma in situ;
13. Anti-tumor therapies within 4 weeks prior to the initiation of investigational treatment, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy and immunotherapy;
14. Palliative radiotherapy for a bone metastasis lesion within 2 weeks prior to the initiation of investigational treatment;
15. Surgery prior to enrolment within 28 days prior to the initiation of investigational treatment or unhealed surgical incision;
16. Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for hair loss);
17. Clinically significant active infection;
18. Human immunodeficiency virus (HIV) infection;
19. History of clinically significant hepatic diseases, including viral hepatitis, (Hepatitis B carriers with active HBV infection, i.e., HBV DNA positive [>1×104/ml]; Hepatitis C virus infection with HBV RNA positive [>1×103/ml]); or other types of hepatitis, and liver cirrhosis.
20. Women who are pregnant or lactating;
21. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of disease stability of longer than 14 days;
22. Inability to orally take medicine, dysphagia or an active gastric ulcer resulting from previous surgery or a severe gastrointestinal disease, or any other condition that investigators believe may affect absorption of the investigational product;
23. Receive investigational treatment in another clinical study within the 4 weeks prior to enrolment;
24. Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may prohibit use of the investigational product, affect interpretation of study results, or put the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AE/SAEs | from day 1 of first dosing to 30 days after permanent discontinuation of Sulfatinib
  the safety of Sulfatinib

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, MD, Study Director — Hutchison Medi Pharma
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - the 307 Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided